CLINICAL TRIAL: NCT04738669
Title: Effectiveness of Mhealth and Teach-back Methods in Readmissions Reduction in Prime Minister's National Health Programme - A Feasibility Randomized Controlled Trial
Brief Title: Mhealth and Teach-Back Effectiveness In 30-Day Readmissions Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Health Services Academy, Islamabad, Pakistan (Other)
Responsible Party: Principal Investigator, Syed Fawad Mashhadi, PhD Fellow, Health Services Academy, Islamabad, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: No 1-07/14-HSA/2021
Record Dates: First submitted 2021-01-21; First posted 2021-02-04 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Readmission; mHealth; Teach-Back Communication
Keywords: Readmission; Mobile health; mHealth; Teach-Back Communication
MeSH Terms: conditions — Teach-Back Communication | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention): No intervention is being conducted in this arm. Routine care is being given to these patients. The patients will be followed up for any readmissions during the intervention period.
- mHealth Arm (Experimental): This arm will receive first receive weekly telephone call followed by the SMS in Urdu regarding medication adherence according to the discharge instructions.
  The calls and SMS will be sent on 7, 14, 21 and 30th day post-index discharge. The patients will be followed up for any readmissions during the intervention period.
  Interventions: Other: mHealth
- Teach back arm (Experimental): The trained doctors thoroughly explained the discharge instructions, medication schedule and any other self-care instructions to these participants and asked them to repeat what they have understood from the doctor verbal counselling.
  If the instructions were not clearly comprehended by the patients, then the same would be repeated by the consultant doctor.
  The patients will be followed up for any readmissions during the intervention period.
  Interventions: Behavioral: Teach-back

INTERVENTIONS:
Other: mHealth — The mHealth intervention includes telephonic call and SMS.
  Arms: mHealth Arm
Behavioral: Teach-back — While the teach-back includes counselling session related to discharge instruction including medication adherence.
  Arms: Teach back arm

SUMMARY:
The Study is a feasibility randomized controlled trial aiming to assess the feasibility of mHealth (voice call and SMS) and teach-back interventions on reducing the 30 days readmission rate in the patients enrolled in the Sehat Sahulat Programme (Prime Minister National Health Programme(PMNHP)).

The prime objective of this study was to generate a proof of concept for the conduct of a definitive trial for the reduction in readmissions in PMNHP.

A feasibility randomized controlled trial study consisted of three arms i.e intervention 1 (telephonic contact and text messages), intervention 2 (teach-back method) and control is planned in program beneficiaries of Islamabad, Pakistan.

The trial is being carried out in the three hospitals of Islamabad and patients are being recruited as per the inclusion and exclusion criteria.

DETAILED DESCRIPTION:
Interventional Description of intervention(s) / exposure The study will comprise of three phases Phase I = Preparation Phase II= Implementation and monitoring Phase III = Evaluation Phase I (Preparation) i. Permissions

* Ethical approval from Institutional review Board of Health Services Academy Islamabad
* Permission from PMNHP to carry out a feasibility study
* Written consent from doctors and nurses to be enrolled in the teach-back process
* Informed verbal consent from all the selected patients to be enrolled in the PMNHP ii. Situation analysis The cross-sectional study will be conducted at the start of study prior to intervention to provide baseline data on selected variables. The baseline data will include sociodemographic status, diagnosis, comorbidities, length of stay in the hospital for the index admission.

Phase II (Implementation) i) Team building This step shall include recruiting educated individuals for the survey. For this purpose selected PMNHP staff will be recruited for telephonic contact with the patients.

Researcher himself will brief and orient the team on background and objectives, the usefulness of the study and data recording and medication adherence scale to be used in the study, in a one day workshop comprising of one session of 3 hours.

ii) Validation of the Urdu translation of Medication Adherence Questionaire (MAQ) In order to address the validity and reliability of the MAQ translation and back translations of the questionnaire will be carried out. The questionnaire will be pretested on 10 patients by the staff for adaptability in accordance with the WHO guidelines.

iii) Developing text for SMS This shall comprise of developing easy and understandable text for SMS in English and Urdu for medication adherence and timely follow up to be delivered to the patients. For this purpose, Health communication experts and \ public health professionals will be contacted and involved. The developed SMS will be piloted among patients in a similar setting.

iv) Training of Data collectors for telephonic contact Selected PMNHP staff will be trained to contact the patients on their telephones and ask questions regarding their medication adherence and fill up the MAQ. Training sessions will be conducted by the researcher to carry out a telephonic survey and send SMS messages to the selected patients.

v) Training of doctors and nurses on the teach-back process Doctors and nurses from the selected empanelled hospitals will be trained on the teach-back process for better discharge communication with the patients. One day training session will be held in the Health Services academy vi) Assigning tasks and responsibilities All team members will be provided with a work-plan and agreed on responsibilities with timelines, in order to ensure timely and proper implementation of the various phases of the study.

vii) Intervention: Intervention - 1 (mhealth through a telephonic voice call and text messages) Telephonic voice calls for medication adherence using Morisky, Green and Levine (MGL) 4 items validated medication adherence scale at 7, (Baseline) 14, 21 and 30 days post index discharge. MGL is a validated tool for assessment of medication adherence with a Cronbach alpha = 0.61 in a European setting. The instrument will be translated in Urdu language and will be validated for linguistic and cultural adaptation using the following procedure:-

1. Forward translation One translator, preferably a health professional, familiar with the terminology of the area covered by the instrument and with interview skills will be given this task.
2. Expert panel A bilingual (in English and Urdu) expert panel will be convened. The goal in this step will be to identify and resolve the inadequate expressions/concepts of the translation, as well as any discrepancies between the forward translation and the existing or comparable previous versions of the questions if any. The result of this process will produce a complete translated version of the questionnaire
3. Back-translation Using the same approach as that outlined in the first step, the instrument will then be translated back to English by an independent translator who has no knowledge of the questionnaire
4. Pre-testing and cognitive interviewing. Pre-testing will be done on a sample of 10 - 18 patients and other discrepancies will be removed • Weekly Short text messages (SMS) from PMNHP staff will be sent to the enrolled patients about adherence to medication and follow up reminders

Intervention - 2 ( Teach-Back process) Teach-back is a simple mechanism by which a patient's understanding of a concept or topic may be assessed.

Society of Hospital Medicine (US) complete teach-back module will be used to train nurses and doctors of PMNHP empanelled hospitals in ICT in a one-day training session in Health Services Academy. This teach-back process intervention will be utilized in in group 2

viii) Monitoring the process: All steps and activities of the study will be monitored and spot-checked by the researcher Patients in the study will be contacted through telephone randomly in order to ensure that they are receiving teach-back, SMS and telephonic calls regarding medication adherence and follow up.

Phase III: Trial Acceptability

* In-depth Interviews and Focused Group Discussions from stakeholders at all three levels
* Post-intervention exploration of factors influencing implementation of the Interventions with identification of facilitators and barriers faced by stakeholders during the pilot implementation
* This will generate evidence to support up scalability of PMNHP
* Ten individuals from each level through purposive sampling will be selected for subjective perceptions and acceptability of the interventions

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 30 years of age

  * Incident adult cases with index admission in PMNHP
  * Ischemic Heart disease, Myocardial Infarction, Hypertension, Diabetes Mellitus, Bronchial Asthma
  * Patients with a valid mobile number
  * Able to read the SMS in Urdu

Exclusion Criteria:

* Serious mental illness such as schizophrenia,

  * Are unable to use a telephone
  * Are cognitively impaired during hospitalization as diagnosed by the consultant

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Readmission within 7 days post discharge | 7 days post discharge.
  7 Days after discharge, participants were assessed for readmission.
Readmission within 14 days post discharge | 14 days post discharge.
  14 Days after discharge, participants were assessed for readmission.
Readmission within 21 days post discharge | 21 Days post discharge
  21 Days after discharge, participants were assessed for readmission
Readmission within 30 days post discharge | 30 Days post discharge
  30 Days after discharge, participants were assessed for readmission

CONTACTS AND LOCATIONS:
Overall Officials: Assad Hafeez, PhD, Study Director — Health Services Academy, Pakistan
Locations (1):
- Alkhidmat AlRazi Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT04738669/ICF_000.pdf